CLINICAL TRIAL: NCT02344901
Title: ReAl-life Multicentre Survey Evaluating the Status of Stroke Prevention Strategies in Patients With Non-Valvular Atrial Fibrillation in TurKey (RAMSES)
Brief Title: ReAl-life Multicentre Survey Evaluating Stroke Prevention Strategies (RAMSES)
Acronym: RAMSES
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ozcan Basaran, M.D., Muğla Sıtkı Koçman University
Other Study IDs: RAMSES
Record Dates: First submitted 2015-01-18; First posted 2015-01-26 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Thrombotic Stroke; Atrial Fibrillation and Flutter
Keywords: non-valvular atrial fibrillation; stroke prevention; novel oral anticoagulants; warfarin
MeSH Terms: conditions — Thrombotic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- atrial fibrillation patients: >18 year old. Atrial fibrillation patients without mitral stenosis or any prosthesis.

SUMMARY:
The aim of this study is to evaluate the present status of stroke prevention strategies in patients with non-valvular atrial fibrillation (NVAF). Vitamin K antagonists (VKAs) have been the only available oral anticoagulant therapy for decades. Recently novel oral anticoagulants have emerged as an alternative for VKAs. This study is planned to evaluate the epidemiological characteristics, thromboembolic and bleeding risks, stroke prevention strategies and appropriateness of oral anticoagulant use in NVAF patients. Time in therapeutic range (TTR) is going to be calculated as the percent of visits in range (2-3) for warfarin patients. This is a national multicenter observational study in which Turkey is divided into seven regions. A proportional number of patients to the population of every region is planned to be included.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), classified as nonvalvular (NVAF) in the absence of rheumatic mitral stenosis or valvular prosthesis,is the most common arrhythmia, with an estimated prevalence of 1.5-2%. AF is associated with a greater risk of arterial thromboembolic events, especially cerebrovascular, whose incidence is 5-7 times higher. The risk of death is also doubled, and AF has a greater degree of disability and probability of recurrence than stroke due to other causes. To prevent stroke in patients with NVAF, antithrombotic treatments are employed with oral anticoagulants such as vitamin K antagonists (VKA) and, in a number of circumstances, antiplatelet agents. Although VKA (mainly warfarin) are highly effective to reduce the risk of stroke, and have been the sole choice for stroke prevention during the last 50 years, their use is limited for a number of reasons: narrow therapeutic range, drug and food interactions, need for monitoring, and risk of bleeding. Recently, new oral anticoagulants (NOACs) have been marketed for this indication. The aim of this study was to determine the standard clinical practice followed in the treatment to prevent stroke in patients with NVAF in Turkey. The purpose of this study is to demonstrate the current status of the clinical background of AF patients and to follow, analyze and evaluate patients with AF in a large multicenter nation-wide trial. The primary inclusion criteria will be age ≥18 years and with electrocardiographically confirmed NVAF (eg, by electrocardiogram, Holter monitoring, etc). The enrollment of patients will be started in February 2014. All the participating institutions will enroll all consecutive patients with NVAF under regular outpatient care or under admission.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation

Exclusion Criteria:

* Valvular heart disease (mitral stenosis, prosthetic heart valves, heart valve surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-valvular atrial fibrillaiton patients
Sampling Method: Non-Probability Sample
Enrollment: 6273 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of patients with non-valvular atrial fibrillation receiving appropriate oral anticoagulant for stroke prevention | 2 months

SECONDARY OUTCOMES:
creatinine clearance of patients | 2 months
time in therapeutic range of warfarin using patients | 2 months
CHA2DS2VASc (congestive heart failure or left ventricular dysfunction, hypertension, age ≥75 years, diabetes, thromboembolism or stroke history, vascular disease, age 65-74 years, and sex) score of patients | 2 months
HAS-BLED (hypertension, renal or liver failure, stroke history, bleeding history, labile international normalized ratio, age >65 years, drugs, or alcohol); score of patients | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Murat Biteker, Assoc. Prof., Study Chair — Muğla Sıtkı Koçman University
Locations (62):
- Turkey (Türkiye) (62):
  - Adana Numune Education and Research Hospital, Adana
  - Ankara Kecioren Education and Research Hospital, Ankara
  - Diskapi Yidirim Beyazit Education and Research Hospital, Ankara
  - Medicana International Ankara Hospital, Ankara
  - TOBB ETU Hospital, Ankara
  - Ufuk university Faculty of Medicine, Ankara
  - Antalya Memorial Hospital, Antalya
  - Aydin State Hospital, Aydin
  - Bandirma State Hospital, Balıkesir
  - Gonen State Hospital, Balıkesir
  - Batman State Hospital, Batman
  - Bingol State Hospital, Bingöl
  - Burdur State Hospital, Burdur
  - Iskilip State Hospital, Çorum
  - Diyarbakir Gazi Yasargil Education and Research Hospital, Diyarbakır
  - Elazig Education and Research Hospital, Elâzığ
  - Erzurum Education and Research Hospital, Erzurum
  - Acibadem Eskisehir Hospital, Eskişehir
  - Ersin Arslan State Hospital, Gaziantep
  - Gaziantep 25 Aralik State Hospital, Gaziantep
  - Hatay Iskenderun State Hospital, Hatay
  - Acibadem Kadikoy Hospital, Istanbul
  - Bagcilar Education and Research Hospital, Istanbul
  - Haydarpasa Numune Education and Research Hospital, Istanbul
  - Istanbul Acibadem Maslak Hospital, Istanbul
  - Istanbul Liv Hospital, Istanbul
  - Istanbul Medipol University Medical Faculty, Istanbul
  - Kartal Kosuyolu Education and Research Hospital, Istanbul
  - Kartal Yavuz Selim State Hospital, Istanbul
  - Sisli Etfal Education and Research Hospital, Istanbul
  - Siyami Ersek Education and Research Hospital, Istanbul
  - Sureyyapasa Education and Research Hospital, Istanbul
  - Tuzla State Hospital, Istanbul
  - Gaziemir State Hospital, Izmir
  - Izmir Medical Park Hospital, Izmir
  - Kahramanmaras Necip Fazil Hospital, Kahramanmaraş
  - Kafkas University Medical Faculty, Kars
  - Gebze Fatih State Hospital, Kocaeli
  - Kocaeli Derince Education and Research Hospital, Kocaeli
  - Kocaeli State Hospital, Kocaeli
  - Mevlana University Faculty of Medicine, Konya
  - DPU Evliya Celebi Education and Research Hsopital, Kütahya
  - Luleburgaz State Hospital, Kırklareli
  - Malatya State Hospital, Malatya
  - Mersin Dogus Hospital, Mersin
  - Mersin State Hospital, Mersin
  - Mersin Tarsus State Hospital, Mersin
  - Mersin Toros State Hospital, Mersin
  - Mersin University Medical Faculty, Mersin
  - Mut State Hospital, Mersin
  - Fethiye State Hsopital, Muğla
  - Mugla Sitki Kocman University Education and Research Hospital, Muğla
  - Samsun Education and Research Hospital, Samsun
  - Samsun Medical Park Hospital, Samsun
  - Sanliurfa Balikligol State Hospital, Sanliurfa
  - Suruc State Hospital, Sanliurfa
  - Sivas Cumhuriyet University Medical Faculty, Sivas
  - Sivas Numune State Hospital, Sivas
  - Gaziosmanpasa University Medical Faculty, Tokat Province
  - Trabzon Ahi Evren Education and Research Hospital, Trabzon
  - Usak State Hospital, Uşak
  - Yozgat State Hospital, Yozgat

REFERENCES:
- [Derived] Mert KU, Mert GO, Basaran O, Beton O, Dogan V, Tekinalp M, Aykan AC, Kalaycioglu E, Bolat I, Tasar O, Safak O, Kalcik M, Yaman M, Kirma C, Biteker M; RAMSES investigators. Real-world stroke prevention strategies in nonvalvular atrial fibrillation in patients with renal impairment. Eur J Clin Invest. 2017 Jun;47(6):428-438. doi: 10.1111/eci.12758. Epub 2017 May 16. PMID 28407216
- [Derived] Biteker M, Basaran O, Dogan V, Altun I, Ozpamuk Karadeniz F, Tekkesin AI, Cakilli Y, Turkkan C, Hamidi M, Demir V, Gursoy MO, Tek Ozturk M, Aksan G, Seyis S, Balli M, Alici MH, Bozyel S. Real-World Clinical Characteristics and Treatment Patterns of Individuals Aged 80 and Older with Nonvalvular Atrial Fibrillation: Results from the ReAl-life Multicenter Survey Evaluating Stroke Study. J Am Geriatr Soc. 2017 Aug;65(8):1684-1690. doi: 10.1111/jgs.14855. Epub 2017 Apr 10. PMID 28394435
- [Derived] Basaran O, Dogan V, Beton O, Tekinalp M, Aykan AC, Kalaycioglu E, Bolat I, Tasar O, Safak O, Kalcik M, Yaman M, Inci S, Altintas B, Kalkan S, Kirma C, Biteker M; and Collaborators. Impact of valvular heart disease on oral anticoagulant therapy in non-valvular atrial fibrillation: results from the RAMSES study. J Thromb Thrombolysis. 2017 Feb;43(2):157-165. doi: 10.1007/s11239-016-1445-1. PMID 27848065
- [Derived] Basaran O, Beton O, Dogan V, Tekinalp M, Aykan AC, Kalaycioglu E, Bolat I, Tasar O, Safak O, Kalcik M, Yaman M, Altun I, Soylu MO, Kirma C, Biteker M; RAMSES Study. ReAl-life Multicenter Survey Evaluating Stroke prevention strategies in non-valvular atrial fibrillation (RAMSES study). Anatol J Cardiol. 2016 Oct;16(10):734-741. doi: 10.14744/AnatolJCardiol.2016.6752. PMID 27723665
- [Derived] Basaran O, Dogan V, Beton O, Tekinalp M, Aykan AC, Kalaycioglu E, Bolat I, Tasar O, Safak O, Kalcik M, Yaman M, Inci S, Altintas B, Kalkan S, Kirma C, Biteker M; and Collaborators. Suboptimal use of non-vitamin K antagonist oral anticoagulants: Results from the RAMSES study. Medicine (Baltimore). 2016 Aug;95(35):e4672. doi: 10.1097/MD.0000000000004672. PMID 27583892
- [Derived] Basaran O, Dogan V, Memic Sancar K, Altun I, Mert KU, Mert GO, Basaran NF, Cekic EG, Kirma C, Biteker M; RAMSES investigators. Rationale, design and methodology of the RAMSES Study: ReAl-life Multicenter Survey Evaluating Stroke Prevention Strategies. Turk Kardiyol Dern Ars. 2016 Apr;44(3):215-20. doi: 10.5543/tkda.2015.29266. PMID 27138310